CLINICAL TRIAL: NCT05048459
Title: Randomized Clinical Trial of Tele-Surveillance and Remote Symptom Monitoring Compared to Standard Surveillance for HPV-Associated Oropharynx Cancer With No Evidence of Disease on Post-Treatment Imaging
Brief Title: Comparing Two Surveillance Approaches for People Who Have Received Treatment for HPV-associated Head and Neck Cancer and Show No Signs of Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-347
Record Dates: First submitted 2021-09-01; First posted 2021-09-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Squamous Cell Carcinoma
Keywords: Tele-Surveillance; Remote Symptom Monitoring; 21-347; HPV-associated Head and Neck Cancer
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The study design is a 1:1 randomized clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard surveillance (Active Comparator): This surveillance approach involves the participant coming to the clinic for in-person follow-up visits and having routine endoscopy and cancer imaging procedures as needed
  Interventions: Other: Standard surveillance; Other: Questionnaires
- Telemedicine surveillance (tele-surveillance) (Experimental): Tele-surveillance involves the participant staying at home while their healthcare providers follow their condition and give them the care they need. They can communicate with their healthcare team through face-to-face video conferencing on their desktop computer, laptop, smart phone, or tablet. They can also communicate with their healthcare team by phone.
  Interventions: Other: Telemedicine surveillance (tele-surveillance); Other: Questionnaires

INTERVENTIONS:
Other: Standard surveillance — Participant coming to the clinic for in-person follow-up visits and having routine endoscopy and cancer imaging procedures as needed
  Arms: Standard surveillance
Other: Telemedicine surveillance (tele-surveillance) — The tele-surveillance visit occurs annually after completion of therapy and consists of a phone call with or without video conferencing between the patient and the treatment team (physician, nurse, and/ or nurse practitioner). The use of video conferencing is strongly encouraged. Clinic visits, endoscopies, and imaging studies can be performed at the discretion of the treatment team for concerning patient symptoms.
  Arms: Telemedicine surveillance (tele-surveillance)
Other: Questionnaires — EORTC QLQ-C30 and EORTC QLQ-HN43 at 12 and 24 months, FACE-Questionnaire Module, Telehealth Usability Questionnaire, Telehealth Usability Questionnaire, Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction -Patient Satisfaction inventory

SUMMARY:
The purpose of this study is to compare standard surveillance with telemedicine surveillance (tele-surveillance) and find out which surveillance approach is best for people with HPV-associated head and neck cancer who have no evidence of disease after treatment. The researches will look at how the two approaches affect participants' quality of life, health outcomes, and expenses (for example, costs of routine visits and procedures). They will also determine doctors' and patients' satisfaction with tele-surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* ECOG 0-3
* Pathologically (histologically or cytologically) diagnosis of HPV associated squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or oropharyngeal walls)
* No evidence of disease on post-treatment PET/CT within 9 months of completing radiation therapy. No evidence of disease is a consensus determination by the patient's radiation, medical, and surgical oncologist. If the first PET/CT is equivocal, then a second PET/CT can be obtained within 9 months of completing radiation therapy.
* Post-treatment diagnostic imaging with either CT or MRI (recommended but not required)
* Able to speak and read English fluently
* Able to provide informed consent

Exclusion Criteria:

* Patients on clinical trials related to head and neck cancer that have protocol defined follow up activities
* Incomplete response or recurrent disease on post-treatment PET/CT
* Completion of radiation and chemotherapy more than 9 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  PFS will be defined as pathologic evidence of local or distant tumor progression or death from any cause. Patients

SECONDARY OUTCOMES:
Locoregional recurrence (LRR) | 2 years
  Any pathologic evidence of tumor progression in the head and neck will be counted as a LRR. Patients without concerning symptoms as determined by the treating physician at the time of the tele-visit will be determined to be free of LRR. If imaging or biopsies or ordered at any time and are consistent with tumor progression, then these patients will be counted as having a LRR event. both the EORTC QLQ-C30 and EORTC QLQ-HN43 Scores of all scales and single-item measures range from 0 to 100 with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm